CLINICAL TRIAL: NCT00471692
Title: A Randomised, Double Blind, Placebo Controlled Study to Compare Ilio Inguinal Nerve Block and Local Wound Irrigation
Brief Title: Local Anaesthetic Following Hernia Repair
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to high incidence of neurological complication in those with ilioinguinal block
Sponsor: Royal Hobart Hospital (Other Government)
Responsible Party: Principal Investigator, Stuart Walker, Staff Specialist, Royal Hobart Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H0008762
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Inguinal Hernias
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Normal saline placebo
  Interventions: Drug: Ropivicaine
- Ropivocaine (Active Comparator): Ilioinguinal nerve block with ropivocaine
  Interventions: Drug: Ropivicaine

INTERVENTIONS:
Drug: Ropivicaine

SUMMARY:
Inguinal hernia repair is a common surgical procedure. The major current debates revolve around laparoscopic hernia repair. The most recent Cochrane review concluded that laparoscopic inguinal hernia repair was associated with less post operative and chronic pain, shorter convalescence and earlier return to work when compared to open repair (McCormack K, Scott NW, Go PM, Ross S, Grant AM. EU hernia trialist collaboration. Laparoscopic techniques versus open techniques for inguinal hernia repair. Cochrane Database Syst Rev 2003; 1(CD001785.). However, laparoscopic repair has not gained wide acceptance. It is more expensive, technically difficult for the inexperienced surgeon, is associated with rare but potentially more hazardous procedure related complications (Lo CH, Trotter D, Grossberg P. Unusual complications of laparoscopic totally extraperitoneal inguinal hernia repair. ANZ journal of Surgery 2005 Oct, 75(10): 917 - 919.) and unlike open repair, requires a general anaesthetic. Critics state that laparoscopic repair is not suitable for all general surgeons and should be restricted to experts. Two prospective studies have shown that a longer laparoscopic learning curve exists when compared to open surgery. Up to 200 laparoscopic procedures are required to achieve a recurrence rate comparable to open mesh repair. (Bittner R, Schmedt CG, Schwarz J, Kraft K, Leigl BJ. Laparoscopic transperitoneal procedure for routine repair of groin hernia British journal of Surgery 2002 89; 1062 - 1066.) A meta-analysis and large multicentre randomised study have added to these concerns by demonstrating a higher recurrence rate with laparoscopic repair. (Memon MA, Cooper NJ, Memon B, Memon MI, Abrams KR. Meta-analysis of randomised controlled trials comparing open and laparoscopic inguinal hernia repair. British journal of Surgery 2003; 90: 1479 - 1492. Neumayer L, Giobbie-Hurder, Jonasson O, Fitzgibbons R, Dunlop D, Gibbs J et al. Open mesh versus laparoscopic mesh repair of inguinal hernias. New England Journal of Medicine 2004; 350: 1819 - 1827.). Over the period 1998 to 2003, in Denmark, the frequency of laparoscopic repair remained constant at 4.5 - 8.0%, the laparoscopic approach being used more frequently for bilateral hernia repairs and recurrent hernia repairs. There was a higher re-operation rate following laparoscopic repair of bilateral inguinal hernias compared to bilateral open hernia repair. (Wara P, Bay-Nielsen M, Juul P, bendix J, Kehlet H. Prospective nationwide analysis of laparoscopic versus Lichenstein repair of inguinal hernia. British Journal of Surgery 2005 92(10); 1277 - 1281.)

Given these issues, a considerable number of adult inguinal hernia repairs will continue to be performed using the open technique. There is the opportunity to improve the results of open repair by potentially improving post operative pain and chronic pain. One method may be to perform an ilio inguinal nerve block. However, this procedure can be complicated by femoral nerve palsy, colonic or small bowel puncture and pelvic haematomas (Johr M, Sossai R. Colonic puncture during ilioinguinal nerve block in a child. Anesth Analg 1999 88 1051 - 1052, Amory C, mariscal A, Guyot E et al. Is ilioinguinal/iliohypogastric nerve block always totally safe in children? Paediatr Anaesth 2003; 13: 164 - 166. Vaisman J. Pelvic hematoma after an ilioinguinal nerve block for orchialgia Anesth Analg 2001 92 1048 - 1049. Notaras MJ. Transient femoral nerve palsy complicating preoperative ilioinguinal nerve blockade for inguinal herniorrhaphy. British Journal of Surgery 1995 82: 854. Rosario DJ, Skinner PP, Raftery AT. Transient femoral nerve palsy complicating preoperative ilioinguinal nerve blockade for inguinal herniorrhaphy. British journal of Surgery 1994 81: 897. Ghani KR, McMillan R, Paterson-Brown S. Transient femoral nerve palsy following ilio-inguinal nerve blockade for day case inguinal hernia repair. J R Coll Surg Edinb 2002; 47: 626 - 629. Erez I, Buchumensky V, Shenhman Z, et al. Quadriceps paresis in pediatric groin surgery. Pediatr Surg Int 2002; 18: 157 - 158, Vironen J, Neiminen J, Eklund A, Paavolainen P. Randomised clinical trial of Lichtenstein patch or prolene hernia system for inguinal hernia repair. British Journal of Surgery 2006; 93: 33 - 39)), resulting in delayed discharge of patients. It also has a failure rate of 20 - 30% (Lim SL, Ng SB, Tan GM. Ilioinguinal and iliohypogastric nerve block revisited; single shot versus double shot technique for hernia repair in children. Paediatr Anaesth 2002; 12; 255 - 260.) The aim of our study is therefore to assess the role of ilio inguinal nerve block in adult patients undergoing primary inguinal hernia repair.

DETAILED DESCRIPTION:
Patients presenting to the Royal Hobart Hospital for open surgery to an inguinal hernia were approached for inclusion to the study. To patient refused entry. Informed consent was obtained and the study was approved by the local ethics and research committees.

Following induction of general anaesthesia, a sealed envelop was opened. This envelop was prepared by the pharmacy department at the Royal Hobart Hospital. This envelope contained two syringes presented sterile, each containing a clear liquid. The syringe labelled ilioinguinal nerve block was given to the anaesthetist for insertion of an "ilioinguinal nerve block" prior to surgical preparation and draping. The second syringe, labelled wound infiltration was given to the scrub nurse for wound irrigation by the surgeon prior to closure of the external oblique aponeurosis. Patients were divided into the following groups:

Group 1 - 20mls 0.5% ropivacaine for ilio inguinal nerve block and 20mls saline for wound irrigation.

Group 2 - 20mls saline for ilioinguinal nerve block by anaesthetist and 20ml ropivacaine 0.5% for wound irrigation

Group 3 - 20mls saline for ilioinguinal nerve block and 20mls saline for wound irrigation.

GA protocol:

* 0.03mg/kg midazolam IV
* 2mcg/kg fentanyl
* Propofol to induce anaesthesia
* Laryngeal mask.
* Maintenance with oxygen/air and sevoflurane
* Dexamethasone 8mg IV for prophylaxis of post operative nausea and vomiting
* 100mg PR diclofenac
* 1g IV paracetamol

Technique for ilioinguinal nerve block:

Puncture site 1cm medial to anterior superior iliac spine and a fascial click is detected before injection of local anaesthetic. i.e. just below external oblique.

All patients were prescribed a fentanyl PCA for 2 hours postoperatively (1000mcg in 50ml normal saline with a bolus dose of 25mcg set for every 3 minutes. No background rate. If the patient was unable to press the button, nursing staff did this until the patient was able to do so). Using the PCA machine we were be able to record the number of PCA requests and the total PCA fentanyl delivered.

Post operative outcome measures. On an hourly basis until discharge, patients were asked to rate their pain as none, mild, moderate or severe. They were also presented with a visual analogue scale for post operative pain.

On day one, two, fourteen and twenty eight post operatively, the patient was telephoned at home and asked to grade their pain on a scale of none, mild, moderate or severe for:

* On going to bed at night
* The worst pain they had overnight
* Getting out of bed in the morning.

Amount of post operative analgesia required will be asked at the time of the telephone call.

Patients were also asked for the time for return to:

* Walking without discomfort
* Exercise without discomfort
* Sexual activity
* Work

All operations were performed by the same consultant surgeon or by a surgical registrar under direct supervision of the consultant surgeon. All patients had a standard prolene mesh repair.

Primary end point. Post operative analgesia requirements. Visual analogue scores.

Secondary end points. Return to normal activities.

Statistics. For an 80% chance of detecting a difference in visual analogue scale with standard deviation of 0.5 and p<0.05, 30 patients would be required in each group.

ELIGIBILITY:
Inclusion criteria:

* Primary unilateral inguinal hernia
* Aged 18 years or more

Exclusion criteria:

* Bilateral inguinal hernia repairs to be performed at the same procedure.
* Recurrent inguinal hernia
* Patient unable to give informed consent
* Contraindication to the use of local anaesthetic
* Operation to be performed under local or spinal anaesthetic.
* Contraindication to use of diclofenac, fentanyl or paracetamol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Post operative analgesia requirements. Visual analogue scores. | Hourly following surgery

SECONDARY OUTCOMES:
Return to normal activities. | 4 weeks post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Stuart walker, Principal Investigator — Royal Hobart Hospital
Locations (1):
- Royal Hobart Hospital, Hobart, Tasmania, Australia